CLINICAL TRIAL: NCT03675256
Title: KENya Single-dose HPV-vaccine Efficacy - The KEN-SHE Study
Brief Title: The KEN SHE Study on HPV-vaccine Efficacy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Ruanne Barnabas, MBChB, MSc, DPhil., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022P001178; OPP1188693 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2018-09-06; First posted 2018-09-18 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: At the start of our study, young women will be randomly sorted into three arms. In arm 1, the women will receive the bivalent HPV vaccine. In arm 2, the women will receive the nonavalent HPV vaccine. And in arm 3, the women will receive a meningococcal vaccine. At the crossover vaccine timepoint, those in arms 1 and 2 will receive the meningococcal vaccine, while those in arm 3 will receive either the bivalent or nonavalent HPV vaccine. The three arm study structure makes it possible to compare the women who received an HPV vaccine to those who did not receive an HPV vaccine during the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is blinded. The pharmacists, unblinded data manager, and unblinded statistician are the only ones who will know treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): immediate Cervarix, delayed MenVeo vaccine
  Interventions: Biological: immediate Cervarix, delayed MenVeo vaccine
- Arm 2 (Experimental): immediate Gardasil 9, delayed MenVeo vaccine
  Interventions: Biological: immediate Gardasil 9, delayed MenVeo vaccine
- Arm 3 (Active Comparator): immediate MenVeo, delayed Gardasil 9 vaccine
  Interventions: Biological: immediate MenVeo vaccine, delayed Gardasil 9

INTERVENTIONS:
Biological: immediate Gardasil 9, delayed MenVeo vaccine — Intervention is immediate administration of 9-valent HPV vaccine and delayed MenVeo vaccine
  Arms: Arm 2
Biological: immediate MenVeo vaccine, delayed Gardasil 9 — Intervention is immediate administration of MenVeo vaccine and delayed administration of Gardasil 9
  Arms: Arm 3
Biological: immediate Cervarix, delayed MenVeo vaccine — Intervention is immediate administration of bivalent HPV vaccine and delayed MenVeo vaccine
  Arms: Arm 1

SUMMARY:
The KEN SHE Study aims to identify effective cervical cancer prevention strategies. Cervical cancer is caused by an infection with Human Papillomavirus, also called HPV. In Kenya, about 2,500 women die from this condition each year. The study is conducted by Kenya Medical Research Institute (KEMRI) sites, based in Kisumu, Thika and Nairobi and the University of Washington, Seattle, USA.

The purpose of this study is to learn whether a single dose of the HPV vaccine prevents HPV infection among adolescents and young women. Using a single dose will lower the cost of providing HPV vaccination (compared to two doses) and will make it possible for more women to receive the vaccination and be protected from cervical cancer.

The study will involve approximately 21 clinic visits over a period of 55 months. All visits will involve blood draws and many will involve pelvic swabs. Participants will receive an FDA-approved HPV vaccine and a meningococcal vaccine.

DETAILED DESCRIPTION:
Cervical cancer is the leading cause of new cancer cases among women in Africa. Preliminary evidence suggested a single-dose of the HPV vaccine would be over 95% effective in preventing vaccine type-specific HIV infection, supporting HPV vaccination as a scaleable intervention for cervical cancer prevention. The overall aim of the study is to provide timely results of both single-dose HPV vaccine efficacy and estimates of the cost, cost-effectiveness, and budget impact for dissemination and translation to policy. Several HPV vaccines are available. The KEN SHE Study will determine the efficacy of two HPV vaccines: bivalent and nonavalent vaccines.

At the start of the study, young women were randomly sorted into three arms. In arm 1, the women received the bivalent HPV vaccine. In arm 2, the women received the nonavalent HPV vaccine. And in arm 3, the women received a meningococcal vaccine. The three-arm study structure makes it possible to compare the women who received an HPV vaccine to those who did not receive an HPV vaccine during the study. A formal primary analysis was planned to be conducted after 18 months of follow-up to provide early evidence on single-dose HPV vaccine efficacy.

The principal results of the primary analysis conducted 18 months after enrollment were to demonstrate whether the single-dose HPV vaccine strategy prevents incident persistent HPV vaccine type specific infection among young women, by comparing the rate of new HPV infections among women who receive the vaccine immediately to those receiving delayed vaccination. Single dose HPV vaccination was highly effective at the month 18 primary analysis timepoint. Thus, as recommended by the Data Saftey Monitoring Board, participants should receive a blinded crossover vaccination. Participants who received the HPV vaccine at enrollment will receive the meningococcal vaccine and participants who received the meningococcal vaccine at enrollment, will receive the HPV vaccine (i.e. crossover vaccination). Questions remain regarding the durability of single-dose HPV vaccine efficacy which may limit the uptake of single-dose HPV vaccination. To ensure that vaccine efficacy is durable, crossover vaccination and follow-up will be conducted using a blinded crossover study design. This design will allow comparison of the early and late vaccine efficacy to ensure that single-dose HPV vaccine clinical efficacy does not wane over time. Thus, the study will contribute data on both single-dose HPV vaccine efficacy and durability of the effect. A final analysis will be conducted with the conclusion of up to 55 months of follow-up; if waning protection is detected, participants will receive the World Health Organization recommended course of HPV vaccination.

With the introduction of the crossover vaccination, the primary study endpoint is now persistent vaccine type specific HPV infection at months 18 and 18 months after blinded crossover vaccination. The quantitative antibody response will be documented at months 1 and 24 to support immunobridging analyses to girls and adolescents for the single-dose bivalent and nonavalent vaccines. Using the data on persistent infections and health economic models, we will assess the impact on cervical cancer incidence. Specifically, investigators will compare the incidence of high-risk vaccine HPV types overall and the distribution of HPV types by study arm. Investigators will assess the immunologic response to single-dose HPV vaccination, specifically regarding long lasting B cell responses to support the durability of the single-dose vaccination approach. Data on the magnitude of the antibody response at months 1 and 24 will support immunobridging analyses to young girls and adolescents. The 24 month antibody result will be used to assess durability of the response and will be directly comparable to other studies of the single-dose HPV vaccine which are uniformly using the month 24 antibody result as the primary outcome. Further, among the women who received immediate HPV vaccine, investigators will estimated the durability of the bivalent and nonavalent HPV vaccines by measuring the antibody response and cumulative incidence of persistent cervical HPV over the duration of follow-up. Costing analyses will assess the resources required for scale-up of single-dose HPV vaccination.

Enrollment took 12 months and there are 55 months of follow-up for each participant. The endpoint-driven trial design among women at risk of HPV acquisition will provide primary results after 18 months of follow-up, and, with the extended follow-up, evidence on durability over three years. The study duration is 78 months.

ELIGIBILITY:
Inclusion Criteria:

* Born female
* Age 15 to 20 years
* HIV-negative
* No history of HPV vaccination
* Sexually active: history of 1-5 lifetime partners
* Resident within study area without plans to move away in the next 37 months

Exclusion Criteria:

* Allergies to vaccine components or latex,
* Pregnancy
* Hysterectomy
* Autoimmune, degenerative, and genetic diseases
* Investigator discretion

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2275 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Persistent HPV 16/18 infection across arms | Primary analysis at month 18
  Incident persistent HPV 16/18 infection across arms to measure HPV16/18 and HPV 16/18/31/33/45/52/58/6/11 vaccine efficacy
Persistent HPV 16/18/21/33/45/52/58 infection across arms | Primary analysis at month 18
  Incident persistent HPV 16/18/21/33/45/52/58 infection across the HPV 16/18/31/33/45/52/58/6/11 and immediate meningococcal (delayed HPV) vaccine arms to measure HPV 16/18/31/33/45/52/58/6/11 vaccine efficacy
Durability of HPV vaccine efficacy using blinded crossover vaccination design | Primary analysis 18 months after crossover vaccination
  Incident persistent HPV 16/18/21/33/45/52/58 infection will be compared between the early and late vaccine efficacy periods

SECONDARY OUTCOMES:
Non-inferiority of vaccine response in girls aged 15-20 compared to girls age 9-14 | Secondary analysis at 24 months after enrollment and 18 months post crossover vaccination
  Antibody response after single-dose bivalent or nonavalent vaccination in 15-20 year old adolescents compared to 9-14 year old girls in the DoRIS study
Cost of single-dose HPV vaccination | Secondary analysis at 18 months post crossover vaccination
  Cost of single-dose HPV vaccination to support implementation strategies for single-dose HPV vaccination following World Health Organization recommendation in high cervical cancer burden settings.
Cost-effectiveness of single-dose HPV vaccination | Secondary analysis at 18 months post crossover vaccination
  Cost-effectiveness of single-dose HPV vaccination to support implementation strategies for single-dose HPV vaccination following World Health Organization recommendation in high cervical cancer burden settings.
Budget impact of single-dose HPV vaccination | Secondary analysis at 18 months post crossover vaccination
  Budget impact of single-dose HPV vaccination to support implementation strategies for single-dose HPV vaccination following World Health Organization recommendation in high cervical cancer burden settings.
Immune memory following single-dose HPV vaccination | Secondary analysis at 19 months post crossover vaccination
  B-cell marker levels following single-dose bivalent and nonavalent vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Ruanne Barnabas, MBChB, DPhil, Principal Investigator — Massachusetts General Hospital; Nelly Mugo, MBChB, MPH, Principal Investigator — Kenya Medical Research Institute
Locations (3):
- Kenya (3):
  - Partners in Health, Research and Development, Thika, Kiambu County
  - Kargeno Research and Policy Hub, Kisumu, Nyanza
  - Center for Clinical Research, Nairobi

REFERENCES:
- [Derived] Barnabas RV, Brown ER, Onono MA, Bukusi EA, Njoroge B, Winer RL, Galloway DA, Pinder LF, Donnell D, N Wakhungu I, Biwott C, Kimanthi S, Heller KB, Kanjilal DG, Pacella D, Morrison S, A Rechkina E, L Cherne S, Schaafsma TT, McClelland RS, Celum C, Baeten JM, Mugo NR; KEN SHE Study Team. Durability of single-dose HPV vaccination in young Kenyan women: randomized controlled trial 3-year results. Nat Med. 2023 Dec;29(12):3224-3232. doi: 10.1038/s41591-023-02658-0. Epub 2023 Dec 4. PMID 38049621
- [Derived] Barnabas RV, Brown ER, Onono MA, Bukusi EA, Njoroge B, Winer RL, Galloway DA, Pinder LF, Donnell D, Wakhungu I, Congo O, Biwott C, Kimanthi S, Oluoch L, Heller KB, Leingang H, Morrison S, Rechkina E, Cherne S, Schaafsma TT, McClelland RS, Celum C, Baeten JM, Mugo N. Efficacy of single-dose HPV vaccination among young African women. NEJM Evid. 2022 Jun;1(5):EVIDoa2100056. doi: 10.1056/EVIDoa2100056. Epub 2022 Apr 11. PMID 35693874
- [Derived] Barnabas RV, Brown ER, Onono M, Bukusi EA, Njoroge B, Winer RL, Donnell D, Galloway D, Cherne S, Heller K, Leingang H, Morrison S, Rechkina E, McClelland RS, Baeten JM, Celum C, Mugo N; KEN SHE Study Team. Single-dose HPV vaccination efficacy among adolescent girls and young women in Kenya (the KEN SHE Study): study protocol for a randomized controlled trial. Trials. 2021 Sep 27;22(1):661. doi: 10.1186/s13063-021-05608-8. PMID 34579786
- [Derived] Teppler H, Bautista O; Thomas Group; Flores S, McCauley J, Luxembourg A. Design of a Phase III immunogenicity and safety study evaluating two-dose regimens of 9-valent human papillomavirus (9vHPV) vaccine with extended dosing intervals. Contemp Clin Trials. 2021 Jun;105:106403. doi: 10.1016/j.cct.2021.106403. Epub 2021 Apr 12. PMID 33857679
- [Derived] Kreimer AR, Cernuschi T, Rees H, Saslow D, Porras C, Schiller J. Prioritisation of the human papillomavirus vaccine in a time of constrained supply. Lancet Child Adolesc Health. 2020 May;4(5):349-351. doi: 10.1016/S2352-4642(20)30038-9. Epub 2020 Feb 17. No abstract available. PMID 32078808